CLINICAL TRIAL: NCT02285387
Title: Rhythm Control of AF in Patients With Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0728
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhythm control group (Experimental): 1. Start AAD right after evaluating for LA size, EF, LA thrombus, and presence of CAD during anticoagulation
  2. Cardioversion after 1 month
  3. Rhythm FU schedule (2012 ACC/AHA/ESC guidelines)
  4. If AF recur, RFCA
  Interventions: Procedure: Rhythm control
- Rate control group (Active Comparator): 1. No AAD, just anticoagulation
  2. HR control between 60~110bpm (with beta blocker, calcium channel blocker, digoxin)
  3. Without the treatment about antiarrhythmia and rhythm control, deification of rate control, the subject will be drop out for study.
  Interventions: Procedure: Rate control

INTERVENTIONS:
Procedure: Rhythm control — 1. Start AAD right after evaluating for LA size, EF, LA thrombus, and presence of CAD during anticoagulation
  2. Cardioversion after 1 month
  3. Rhythm FU schedule (2012 ACC/AHA/ESC guidelines)
  4. If AF recur, RFCA
  Arms: Rhythm control group
Procedure: Rate control — 1. No AAD, just anticoagulation
  2. HR control between 60~110bpm (with beta blocker, calcium channel blocker, digoxin)
  3. Without the treatment about antiarrhythmia and rhythm control, deification of rate control, the subject will be drop out for study.
  Arms: Rate control group

SUMMARY:
Prospective randomized (rhythm control or rate control) Objective of study

1. To analyze long term outcome of patients with acute stroke with atrial fibrillation according to the rhythm control
2. To analyze recurrence rate of atrial fibrillation or recurrence stroke in patients with acute stroke according to the rhythm control (by antiarrhythmic drug, cardioversion, catheter ablation)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Atrial fibrillation (20~80 years old)
2. patients with Acute stroke within 7 days
3. LA diameter < 55mm
4. patients possible to anticoagulation and anti arrhythmic drug
5. NIHSS score ≤12

Exclusion Criteria:

1. Hemorrhagic transformation
2. Large cerebral lesion or cerebellar lesion (more than 1/3 of MCA area and 1/2 of ACA area, 1/2 of PCA area, 1/2 of cerebellar area)
3. active internal bleeding
4. Impossible to anticoagulation or anti arrhythmic drug
5. Valvular AF (MA> GII, Mechanical valve, Mitral valve replacement)
6. LV ejection fraction < 30%
7. Structural cardiac disease
8. Catheter ablation history for AF, Cardiac surgery
9. Already prescribed anti arrhythmic drugs
10. With severe medical disease
11. Expected survival < 1year
12. Severe alcoholics, drug addiction

14. Contraindication to MRI 15. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
acute stroke with AF | 1 year
  Long term outcome of rhythm control in patients with acute stroke with AF related to all cause morality, hospital admission, recurrence rate of stroke, major adverse cardiac events
recurrence of silence stroke | 1 year
  Adverse events after anticoagulation or anti arrhythmic drug, recurrence rate after RFCA on AF in patients with stroke, adverse events after RFCA, recurrence rate of silence stroke or clinical stroke
recurrence of AF after rhythm control | 1 year
  Adverse events after anticoagulation or anti arrhythmic drug, recurrence rate after RFCA on AF in patients with stroke, adverse events after RFCA, recurrence rate of silence stroke or clinical stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Park J, Shim J, Lee JM, Park JK, Heo J, Chang Y, Song TJ, Kim DH, Lee HA, Yu HT, Kim TH, Uhm JS, Kim YD, Nam HS, Joung B, Lee MH, Heo JH, Pak HN; RAFAS Investigators*. Risks and Benefits of Early Rhythm Control in Patients With Acute Strokes and Atrial Fibrillation: A Multicenter, Prospective, Randomized Study (the RAFAS Trial). J Am Heart Assoc. 2022 Feb;11(3):e023391. doi: 10.1161/JAHA.121.023391. Epub 2022 Jan 19. PMID 35043663